CLINICAL TRIAL: NCT02845934
Title: Prospective Evaluation of a New Molecular Tool for Early Diagnosis of Mucormycosis
Acronym: MODIMUCOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: N/2013/65
Record Dates: First submitted 2016-07-20; First posted 2016-07-27 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2017-10

CONDITIONS: Mucormycosis
MeSH Terms: conditions — Mucormycosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mucormycosis (Experimental): blood sample
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — additional sampling of blood (estimated volume 6 mL for each sampling) on day of suspicion of the mucormycosis and then twice a week up to a maximum of 8 weeks.

SUMMARY:
This Study evaluates the performance (sensitivity, specificity, positive and negative predictive value values and likelihood ratios) of the DNA detection test for the diagnosis of mucormycosis by comparing it to the routine tests such as CT scan aspects, histopathology, microscopy and fungal culture, in a test group of 52 patients including :

* patients at high-risk according to the EORTC/MSG criteria (patients with prolonged severe neutropenia, receiving corticosteroids or T-cell suppressors, recipients of allogeneic HSCT, or inherited severe immunodeficiency),
* patients with other predisposing factors of invasive mould disease ( diabetes, AIDS, haematological malignancies or solid tumours, trauma, burns); Patients already diagnosed with probable or proven mucormycosis irrespective of underlying conditions.

DETAILED DESCRIPTION:
The patients eligible for this study will already be hospitalized with repeated monitoring of clinical and biological parameters.

Participation in the study will result in an additional sampling of blood (estimated volume 6 mL for each sampling) on day of suspicion of the mucormycosis and then twice a week up to a maximum of 8 weeks.

vials will be added to the routine sampling of these patients (ie, at the time of routine sampling for galactomannan antigemia), and no new sampling procedure will be required.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of invasive mould infection

  * in a patient at high risk according to the EORTC/MSG criteria updated in 2008 (patients with prolonged severe neutropenia, receiving corticosteroids or T-cell suppressor, recipients of allogeneic HSCT, or inherited severe immunodeficiency)
  * or in a patient with other predisposing factors of invasive mould disease ( diabetes, AIDS, haematological malignancies or solid tumours, trauma, burns).
* Patients already diagnosed with probable or proven mucormycosis irrespective of underlying conditions, including patients referred from other centers.
* Only adult patients (18 years or older) will be included

Exclusion Criteria:

* Age : under 18 years
* Patients previously included in the trial with a diagnosis of mucormycosis. However patients previously entered in the trial with a diagnosis other than mucormycosis will be eligible for re- new inclusion.
* Presence of any medical condition that would not allow collection of blood samples for the qPCR test.
* History of documented, successfully treated, prior mucormycosis.
* protected people (pregnant women, minor, guardianship…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
test performance | 8 weeks
  sensitivity, specificity, positive and negative predictive values and likelihood ratios of the DNA serum detection test will be calculated in probable and proven mucormycosis.

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Centre Hospitalier Universitaire, Amiens
  - Centre Hospitalier Régional Universitaire, Besançon
  - AP-HP_Henri-Mondor, Créteil
  - CHU, Dijon
  - HCL, Lyon
  - CHRU, Nancy
  - CHU, Nantes
  - AP-HP_ Necker, Paris
  - AP-HP_St-Louis, Paris
  - CHU, Strasbourg

IPD SHARING:
Plan to Share IPD: No